CLINICAL TRIAL: NCT04271371
Title: Preventing Relapse to Smoking Among Prisoners After Release: Developing and Piloting a Complex Health Intervention
Brief Title: Preventing Relapse to Smoking Among Prisoners After Release
Acronym: PROSPER
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Her Majesty's Prison and Probation Service (HMPPS) (Unknown); Public Health England (Other Government); Cancer Research UK (Other); Plymouth University Peninsula Schools of Medicine & Dentistry (PUPSMD) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 254028
Record Dates: First submitted 2019-09-06; First posted 2020-02-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Smoking; Smoking Reduction; Electronic Cigarette Use
Keywords: Smoking; Smoking Reduction; Electronic Cigarette Use; Prison
MeSH Terms: conditions — Smoking; Smoking Reduction; Vaping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prototype intervention: To be developed through Phase 1 and 2
  Interventions: Other: Not yet developed

INTERVENTIONS:
Other: Not yet developed — A prototype intervention will be developed over Phase 1 & 2 and piloted in Phase 3 of this study.

SUMMARY:
Prisoners experience huge health inequalities, and their exceptionally high smoking prevalence (five times the national average) contributes significantly to their high mortality. Since the introduction of smoke-free polices across Her Majesty's Prison and Probation Service (HMPPS) in England and Wales, prisoners are now obliged to abstain from smoking while held in prison. This represents a unique opportunity to promote lifelong cessation in this highly disadvantaged and marginalised group. However, evidence suggests most prisoners intend to resume smoking as soon as possible after release. A systematic review of prison smoke-free polices worldwide concluded that there was a need for new research to identify effective strategies to reduce relapse in these individuals.

DETAILED DESCRIPTION:
The primary objective of this study will be to develop and pilot test the feasibility and acceptability of an intervention to help prevent prisoners relapse to smoking after release. The study will work in accordance with the Medical Research Council (MRC) framework for developing and evaluating complex interventions. The Preventing Relapse tO Smoking among PrisonErs after Release (PROSPER) study consists of three key Phases:

1. Document the support provided to manage nicotine addiction during imprisonment and in the periods immediately before and after release; establish the extent to which prisoners intentionally resume or unintentionally relapse to smoking after release; and obtain views on how relapse might be prevented.
2. Drawing on current literature and findings from Phase 1, develop and design an prototype intervention to prevent smoking relapse after release.
3. To pilot the designed prototype intervention and conduct a process evaluation to inform the development of further work in this area.

The research will be carried out in three prisons in the East Midlands. The main duties will include recruitment of participants (HMPPS staff members and prisoners), data collection, data analysis, assist with intervention development and refining related intervention materials/resources, co-facilitate Patient and Public Involvement (PPI) groups, contribute to the ethical application for the pilot intervention, and preparation of manuscripts for peer-review publication.

ELIGIBILITY:
Inclusion criteria 2. Release prisoner cohort

* All participants are aged 18 or over (no upper age limit)
* Are currently residing in one of the three study sites (HMPs Nottingham, Ranby and Sudbury)
* Male (women will not be held at any of the study sites)
* Have a provisional release date within the next 2 months.
* Are capable of understanding and consenting to the study.
* Remand and sentenced prisoners.
* Who report that they are a current smoker and/or a current smoker prior to entering prison (smoked up to 7 days before entering prison), and/or were in prison (and still on the same sentence) and a current smoker prior to the smoke-free prison policy.

  3. Reception prisoner cross-sectional
* All participants are aged 18 or over (no upper age limit)
* Are currently residing in the open prison study site (HMP Sudbury)
* Male (women will not be held at any of the study sites)
* Have been in the open prison more than two weeks but for less than 3 months.
* Have been transferred from a closed prison.
* Are capable of understanding and consenting to the study.
* Sentenced prisoners.
* Who report that they were a current smoker prior to entering prison (smoked up to 7 days before entering prison), and/or were in prison (and still on the same sentence) and a current smoker prior to the smoke-free prison policy.

Exclusion criteria 2. Release prisoner cohort

* Present a serious risk of harm to the researchers, highlighted in PNOMIS records or by a member of staff.
* Non-smokers.
* Being deported post release.
* Been in prison for less than four weeks.

  3. Reception prisoner cross-sectional
* Present a serious risk of harm to the researchers, highlighted in PNOMIS records or by a member of staff.
* Been in prison for less than 2 weeks.
* Non-smokers.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants recruited from male prison establishments only
Study Population: Male prisoner population
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
To develop and pilot test the feasibility and acceptability of an intervention to help prevent prisoners relapse to smoking after release. | 3 years
  Smoking abstinence rates at 1 week, 1 month and 3 months post release, self-reported.

SECONDARY OUTCOMES:
To document prisoners smoking history to date and levels of nicotine addiction. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
To document the support provided to manage nicotine addiction during imprisonment and in the periods immediately before and after release. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
The impact of smoke-free prison policy on prisoners smoking behaviours. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
To establish the extent to which prisoners intentionally resume or unintentionally relapse to smoking after release (and does their intended behaviour pre-release predict post-release behaviour). | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
To establish the extent to which prisoners relapse to smoking after transfer to an open prison where smoking is permitted in designated areas. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
To obtain views on triggers to smoking after release (and transfer to an open prison) and how relapse might be prevented. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
For those prisoners who return to smoking after release, at what point do they resume smoking (in days). | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
After release do prisoners use cessation pharmacotherapy, electronic cigarettes or NHS SSS support, or any other means of preventing relapse. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
Record and examine other potential predictors (as outlined in the international literature) of relapse to smoking after release from smoke-free prisons, e.g other negative health behaviours. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
For those prisoners who do return to smoking after release, do they smoke less, the same or more as they previously smoked before entering prison/and or before the prison service went smoke-free. | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
Review of methods of recruitment in prison and community follow-up (to feed into future pilot intervention study). | 1 year
  Phase 1 (Scoping stakeholder interviews/Release prisoner cohort/Reception prisoner cross-sectional)
To develop, design, and refine an intervention to prevent smoking relapse after release with input from fellow academics, stakeholders and PPI groups. | 1 year
  Phase 2 (Intervention development)
To develop logic models to map the problem and the prototype intervention. | 1 year
  Phase 2 (Intervention development)
To assess any barriers and facilitators to the developed intervention. | 1 year
  Phase 3 (Intervention pilot & Intervention process evaluation)
To explore any unintended consequences as a result of the intervention. | 1 year
  Phase 3 (Intervention pilot & Intervention process evaluation)
To identify aspects of the intervention and delivery that could be improved. | 1 year
  Phase 3 (Intervention pilot & Intervention process evaluation)
Explore smoking abstinence rates at 1 week, 1 month and 3 months post release, self-reported and CO validated. | 1 year
  Phase 3 (Intervention pilot & Intervention process evaluation)
Explore impact of the intervention on self-reported health, housing, reconviction rates, use of illicit substances in prisoner's post- release. | 1 year
  Phase 3 (Intervention pilot & Intervention process evaluation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, School of Medicine, Nottingham, Please Select, United Kingdom

IPD SHARING:
Plan to Share IPD: No